CLINICAL TRIAL: NCT03513185
Title: The EARLY Validation and Utility of Somatic Symptom Scale CHINA for Assessing Somatic Symptom Disorder in MYOcardial Outpatients of General Hospital (EARLY-MYO-SSS-CN)
Brief Title: Assessment of SSD in Outpatients Using SSS-CN
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SSSCN2018
Record Dates: First submitted 2018-02-01; First posted 2018-05-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Somatization Disorder
Keywords: somatic symptom disorder; the Somatic Symptom Scale-China; mental disorders management
MeSH Terms: conditions — Somatoform Disorders | interventions — flupentixol, melitracen drug combination; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with SSD: Patients are diagnosed with SSD by physician according to DSM-5,and will be treated with Deanxit, SSRI or SRNI on the basis of severity assessment by physician.
  Interventions: Drug: Deanxit, SSRI or SRNI
- Patients with non-SSD: No SSD is diagnosed by physician according to DSM-5

INTERVENTIONS:
Drug: Deanxit, SSRI or SRNI — After recruiting participants and collecting the baseline data, the SSS-CN, PHQ-15, PHQ-9 and GAD-7 questionnaires will be carried out. An independent diagnosis will be made by primary care physician using the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criterion standard. Deanxit, selective serotonin reuptake inhibitors (SSRI) or serotonin-norepinephrine reuptake inhibitors (SNRI) will be selectively prescribed according to the severity category assessed by physician. Two, 6,10 weeks after patients with correspondent medications, a face-to-face interview, telephone interview or mobile-apps survey will be underwent to follow-up using the SSS-CN, PHQ-15, PHQ-9 and GAD-7 checklists.
  Groups: Patients with SSD

SUMMARY:
About 70-80% of patients with somatic symptom disorder (SSD) visit the general medical hospital instead of psychiatric or other mental health settings. The current self-reporting questionnaires are neither sufficiently considering companioned anxiety or depression nor validated for monitor the treatment efficacy of such group. The Somatic Symptom Scale-China (SSS-CN) is developed due to the urging clinical demanding in general hospital. The study aims to investigate whether the SSS-CN could serve as a timely and practical instrument to detect SSD and assess the severity of the disorder.

DETAILED DESCRIPTION:
One of the most common medical conditions seen in general hospital is somatic symptoms disorder (SSD). As the disorder is characterized by the prominent attention to somatic concerns, patients mainly present initially in medical rather than mental health care settings. The fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) is currently the "gold standard" for the diagnosis of SSD, but it is clinically hard to follow. Thus, It is more clinically practical to detect a disorder by self-administered questionnaires, that patients can score symptoms according to their own condition and severity in a short time. However, the current self-reporting questionnaires, such as the Patient Health Questionnaire-9 (PHQ-9), the Generalized Anxiety Disorder Scale-7 (GAD-7), and the Patient Health Questionnaire-15 (PHQ-15) are neither sufficiently considering companioned anxiety or depression nor validated for monitor the treatment efficacy of SSD patients.

The Somatic Symptom Scale-China (SSS-CN) is developed based on DSM-5 to assess SSD, and it is an abbreviated 20-item version of somatic symptoms that can be entirely self-administered by the patient, but its assessment value has not yet been widely tested. The study aims to investigate whether the SSS-CN could serve as a timely and practical instrument to detect SSD and assess the severity of the disorder.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years old;
2. patients who have no previous diagnosed somatic disease;
3. patients without systemic disease that can account the physical discomfort;
4. patients who agree to take the checklists and undertake assessment from a physician.

Exclusion Criteria:

1. patients who have lost their self-assessed abilities or refuse to participate in;
2. patients who have been previously confirmed serious mental disorders, mental retardation or dementia;
3. patients who are taking anti-anxiety agents or anti-depression agents;
4. patients who are unable to complete at least 1 time follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects are enrolled between September 2017 and June 2020 in the internal medicine department of Renji hospital in Shanghai, China.
Sampling Method: Probability Sample
Enrollment: 1863 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The diagnosis accuracy of somatic burden assessment by SSS-CN | Within 24 hours after collecting the scale.
  The primary objectives of this study are to test the diagnosis accuracy of somatic burden assessment by SSS-CN. Investigators expect that somatic symptom disorder assessed by SSS-CN is as accurate as diagnoses made by the DSM-5 criterion standard

SECONDARY OUTCOMES:
The assessment of treatment efficacy by SSS-CN | Two,6,10 weeks after patients with correspondent medications.
  Investigators hypothesize that the SSS-CN is effective in monitoring treatment efficacy of SSD in primary care patients.
The advantage of SSS-CN | Baseline and 2,6,10 weeks after patients with correspondent medications.
  To explore whether SSS-CN is non-inferior compared with PHQ-15.
SSD companioned with anxiety or depression | Baseline and 2,6,10 weeks after patients with correspondent medications.
  To evaluate how often does SSD companioned with anxiety or depression, or at which circumstance does SSD companioned with anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang M, Zhang W, Su X, Gao C, Chen B, Feng Z, Mao J, Pu J. Identifying and measuring the severity of somatic symptom disorder using the Self-reported Somatic Symptom Scale-China (SSS-CN): a research protocol for a diagnostic study. BMJ Open. 2019 Sep 26;9(9):e024290. doi: 10.1136/bmjopen-2018-024290. PMID 31558447